CLINICAL TRIAL: NCT02067078
Title: The Effect of Protracted Saphenous Nerve and Obturator Nerve Block Versus Saphenous Nerve Block Versus Local Infiltration Analgesia on Opioid Consumption, Pain, Block Duration of Action and Mobilization After Total Knee Arthroplasty.
Brief Title: Protracted Effect of Combined Nerve Blocks After Total Knee Arthroplasty
Acronym: Hobsali
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Regionshospitalet Silkeborg (Other)
Responsible Party: Principal Investigator, Charlotte Runge, MD, Regionshospitalet Silkeborg
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2013-005010-36
Record Dates: First submitted 2014-02-16; First posted 2014-02-20 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Total Knee Arthroplasty; Pain; Nerve Blocks
Keywords: nerve block; total knee arthroplasty; saphenous nerve block; obturator nerve block; pain; opioid consumption
MeSH Terms: conditions — Pain | interventions — Dexamethasone; Bupivacaine; Ropivacaine; Ketorolac Tromethamine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Combined saphenous nerve and obturator nerve block (Experimental)
  Interventions: Drug: Dexamethasone 4 mg + Clonidine 75 microgram + Marcaine 90 mg + Adrenaline 90 microgram
- Saphenous nerve block (Experimental)
  Interventions: Drug: Dexamethasone 2 mg + Clonidine 37,5 microgram + Marcaine 45 mg + Adrenaline 45 microgram
- Local infiltration analgesia (Active Comparator)
  Interventions: Drug: Ropivacaine + Toradol + Adrenaline

INTERVENTIONS:
Drug: Dexamethasone 4 mg + Clonidine 75 microgram + Marcaine 90 mg + Adrenaline 90 microgram — Dexamethasone 4 mg Clonidine 75 microgram Marcaine 90 mg Adrenaline 90 microgram
  Arms: Combined saphenous nerve and obturator nerve block
Drug: Dexamethasone 2 mg + Clonidine 37,5 microgram + Marcaine 45 mg + Adrenaline 45 microgram — Dexamethasone 2 mg Clonidine 37,5 microgram Marcaine 45 mg Adrenaline 45 microgram
  Arms: Saphenous nerve block
Drug: Ropivacaine + Toradol + Adrenaline — Ropivacaine 300 mg + Toradol 45 mg + Adrenaline 0,75 mg
  Arms: Local infiltration analgesia

SUMMARY:
Purpose:

The purpose of this study is to evaluate the postoperative analgesic effect of a combined Saphenous nerve block and Obturator nerve block with local infiltration analgesia in the tissue around the knee after surgery with knee replacement. In the combined nerve blocks we use a mixture of Bupivacaine, Adrenaline, Clonidine and Dexamethasone ("protracted mixture") and the local infiltration consist of Ropivacaine, Adrenaline and Toradol. Our hypothesis is that the combined nerve blocks with protracted mixture prolongs block duration, reduces pain and reduces the need for morphine and thus reduce side effects such as nausea, vomiting and lethargy compared to the current treatment with local infiltration analgesia.

Background:

Nerve blocks as analgesic treatment after orthopedic surgery is a recognized and proven procedure. The nerve blocks have the disadvantage that not only do they anesthetize the sensory nerve fibers but also the nerve fibers to the muscles of the leg. The Saphenous nerve block causes only stunning of sensory nerves to the knee region. The Obturator nerve block causes both stunning of the sensory nerves to the knee region and the thighs inward leading muscles, and does not affect the patient's mobilization capacity.

Both blocks are known to be a good addition to the analgesic treatment. Bupivacaine is a well-known local anesthetic. Adrenaline, Clonidine and Dexamethasone have also been used in other studies, in addition to the local anesthetic agent, and has been shown to prolong the effect of the nerve block. Saphenous and Obturator nerve block with all four drugs Bupivacaine, Adrenaline, Clonidine and Dexamethasone has not been systematically investigated in knee replacement surgery, and it is not known whether this method will provide better pain treatment.

Method

The patient can receive one of three treatments, determined randomly:

* A. Saphenous and Obturator nerve block with active anesthetics (Bupivacaine, Adrenaline, Clonidine, Dexamethasone) and local block around the knee joint with placebo medicine (normal saline).
* B. Saphenous block with active anesthetics and both Obturator nerve block and local block around the knee joint with placebo medicine (normal saline).
* C. Both block with placebo medicine (normal saline) and local block around the knee joint with effective local anesthetic.

Neither patient, investigator or staff around the patient will have knowledge of which treatment the patient has received.

The blocks will be injected before the operation and local infiltration around the knee joint will be given by the surgeon during the operation.

ELIGIBILITY:
Inclusion Criteria:

* Age > 50 years
* Patients set to cemented Total knee arthroplasty in spinal block
* Patients who have given written informed consent to participate in the study after having understood the contents of the protocol and limitations fully
* Illness score 1-3

Exclusion Criteria:

* Patients who can not cooperate with the investigation
* Patients who do not understand or speak Danish
* Patients receiving immunosuppressive therapy
* Patients with a treatment-dependent diabetes mellitus
* Patients with known neuropathy in the lower limbs
* Allergy to those drugs used in the study
* Alcohol and / or drug abuse - the investigator's opinion
* Patients who can not tolerate Non steroid analgesic drugs
* Use of strong opioid several times a day (morphine, ketogan, Oxynorm, methadone, fentanyl)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | 1 to 24 hours postoperatively

SECONDARY OUTCOMES:
Opioid consumption | 1 to 48 hours postoperatively
Pain Score by passive flexion of the knee joint from 0-90 degrees | Time 1, 2, 5, 7, 24, 31, 48 hours postoperatively
  numeric rating scale with values from 0 to 10, with 0 being no pain and 10 being the worst pain imaginable
Pain Score at rest | Time 1, 2 , 5, 7 , 24, 31 and 48 hours postoperatively
  Numeric rating scale with values from 0 to 10, with 0 being no pain and 10 being the worst pain imaginable
Patient-reported time to first postoperative breakthrough pain | Time 1 - 48 hours postoperatively
Nausea | Time 1, 2 , 5, 7 , 24, 31 and 48 hours postoperatively .
  numeric rating scale with values from 0 to 10, where 0 is no nausea and 10 being the worst nausea
Vomiting | Number of between 24 hours postoperatively
Ondansetron | Consumption at time 24 hours postoperative
Number of nights with patient-reported sleep disruptions | Time 48 hours postoperatively
Duration of stay in the post anesthesia care unit | 1 - 48 hours postoperatively
Discharge time from the hospital | Time 1 hour to 2 weeks postoperatively
Patient-reported consumption of opioid | From the discharge date from hospital to ambulatory monitoring 2 weeks postoperatively
Quantitative satisfaction of pain | At 2 weeks postoperatively
  By indicating satisfaction score (0-10 ) , where the value 0 = complete dissatisfaction and 10 = complete satisfaction.
Isometric tests of muscle strength in the hip adductors | 1-2 hours preoperatively and again 30 minutes after the application of obturator nerve blockade
  The patient performed 4-10 measurements with a 30 second break in between each measurement. The difference between the highest value for the test before and after blockade construction calculated.
Time at mobilization to walk with or without support in the form of a walker, crutches or caregivers. | Time 1 to 48 hours postoperatively
Timed Up and Go test | 1-2 hours preoperatively, 24 hours and 2 weeks postoperatively
  The patient rise from a chair and walk round 3 metres and sit on the chair again . The time for completion of the test are recorded .
Cumulated Ambulation Score to illustrate the basic level of mobilization | 1-2 hours pre-operatively, during the first postoperative mobilization, and time 24 hours postoperatively
  The patient scores based on 3 gradations according to their ability to mobilize up and in bed, getting up from a chair and walk with or without aids in the form of high walker or crutches
Movement of the knee joint | 1-2 hours preoperatively, 24 hours and 2 weeks postoperatively
  The patient ability to extend and flex in the knee joint are recorded. The tests are performed with a goniometer

CONTACTS AND LOCATIONS:
Locations (1):
- Regional hospital Silkeborg, Silkeborg, Region Midt, Denmark